CLINICAL TRIAL: NCT06380933
Title: The Effects of Receiving Warm Footbath With Lavender Essential Oil on Sleep and Comfort Among Ventilator-Dependent Patients
Brief Title: The Effects of Receiving Warm Footbath With Lavender Essential Oil on Sleep and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B11103008
Record Dates: First submitted 2024-03-27; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Sleep Quality; Comfort
Keywords: respirator-dependent patient; warm water foot baths; lavender essential oil; sleep quality; comfort level; heartbeat; blood pressure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: two-group crossover design trial and block randomly assigns groups after gender stratification. The experimental group first received a foot bath with lavender essential oil at 41-42C warm water for 20 minutes for 3 days, then rested for 3 days, and then received routine care for 3 days; the control group first received routine care for 3 days, then rested for 3 days, and then received lavender essential oil 41-42C warm water foot bath for 20 minutes for 3 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): foot bath with lavender essential oil for 3 days, and then received routine care for 3 days
  Interventions: Other: experimental group
- control group (No Intervention): first received routine care for 3 days, and then received lavender essential oil with foot bath for 3 days

INTERVENTIONS:
Other: experimental group — first received a foot bath with lavender essential oil at 41-42C warm water for 20 minutes for 3 days, then rested for 3 days, and then received routine care for 3 days
  Arms: experimental group

SUMMARY:
Purposes: Describe the background information and clinical characteristics of respirator-dependent patients, verify the sleep and comfort effects of respirator-dependent patients whether or not they receive a lavender essential oil warm water foot bath, and compare changes of the sleep, comfort, heartbeat, and blood pressure in respirator-dependent patients before and after receiving a lavender essential oil warm water foot bath.

DETAILED DESCRIPTION:
Methods: This study is a randomized clinical trial. It adopts a two-group crossover design trial and block randomly assigns groups after gender stratification. The experimental group first received a foot bath with lavender essential oil at 41-42C warm water for 20 minutes for 3 days, then rested for 3 days, and then received routine care for 3 days; the control group first received routine care for 3 days, then rested for 3 days, and then received lavender essential oil 41-42C warm water foot bath for 20 minutes for 3 days. The measurement tools used self-made structured questionnaires, the Richards-Campbell Sleep Questionnaire （RCSQ）, Numerical Rating of Comfort （NRC）, and heartbeat and blood pressure monitors. Data analysis included descriptive statistics, Chi-square and Fisher's exact correction tests, unpaired t tests and repeated measures ANOVA inferential statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been using a ventilator for 21 days or more
* Individuals aged 45 years or older
* Clear consciousness and the ability to compare hands or hold a pen, with proficiency in Mandarin or Taiwanese communication
* Willingness to participate in the study after receiving an explanation of the research purpose

Exclusion Criteria:

* Individuals with severe mental illness
* Those with cognitive impairments
* Severe visual or hearing impairments
* History of lower limb venous thrombosis
* Amputation or inflammation in the lower limbs
* Muscle contractures in the lower limbs
* Peripheral neuropathy
* Allergic history related to essential oils

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Questionnaire | day 1 and implementation of interventions
  0-100mm

SECONDARY OUTCOMES:
Numerical Rating of Comfort | day1and implementation of interventions
  0-10 points

CONTACTS AND LOCATIONS:
Overall Officials: Hsu M L, BSN, Principal Investigator — Tzu Chi Medical Foundation Dalin Tzu Chi Hospital
Locations (1):
- Hsu Mei-Lian, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aghamohammadi V, Salmani R, Ivanbagha R, Effati Daryani F, Nasiri K. Footbath as a safe, simple, and non-pharmacological method to improve sleep quality of menopausal women. Res Nurs Health. 2020 Dec;43(6):621-628. doi: 10.1002/nur.22082. Epub 2020 Oct 28. PMID 33112004